CLINICAL TRIAL: NCT04712864
Title: A Phase 1, First-In-Human, Open-Label, Multicenter, Multicohort Study of CD4-Targeted Chimeric Antigen Receptor T-Cells (CD4- CAR-T) in Subjects With Relapsed or Refractory T-Cell Lymphoma
Brief Title: Study of CD4-Targeted Chimeric Antigen Receptor T-Cells (CD4- CAR-T) in Subjects With Relapsed or Refractory T-Cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Legend Biotech USA Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB1901-TCL-1001
Record Dates: First submitted 2020-12-01; First posted 2021-01-15 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: T-Cell Lymphoma; Peripheral T-Cell Lymphoma Refractory; Cutaneous T-Cell Lymphoma Refractory; Cutaneous T-Cell Lymphoma Recurrent; Peripheral T-Cell Lymphoma Recurrent
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental LB1901 (Experimental): Drug: anti-CD4 CAR T cells anti-CD4 CAR T cells transduced with a lentiviral vector to express CD4 chimeric receptor domain on T cells.
  Interventions: Biological: LB1901

INTERVENTIONS:
Biological: LB1901 — LB1901 - an autologous CD4-targeted CAR-T immunotherapy

SUMMARY:
This is a Phase 1, first-in-human (FIH), open-label, multicenter, study of LB1901 administered to adult subjects with histologically confirmed CD4+ relapsed or refractory Peripheral T-cell lymphoma (PTCL) (PTCL not otherwise specified [PTCL-NOS] and angioimmunoblastic [AITL]), or relapsed or refractory cutaneous T-cell lymphoma (CTCL) (Sézary syndrome [SS] and mycosis fungoides [MF]).

DETAILED DESCRIPTION:
Study Design: This is a Phase 1, first-in-human (FIH), open-label, multicenter, multicohort study of LB1901 administered to adult subjects with histologically confirmed CD4+ relapsed or refractory Peripheral T-cell lymphoma (PTCL) (PTCL not otherwise specified [PTCL-NOS] and angioimmunoblastic [AITL]), or relapsed or refractory cutaneous T-cell lymphoma (CTCL) (Sézary syndrome [SS] and mycosis fungoides [MF]).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Subjects ≥ 18 years of age.
3. Histologically confirmed diagnosis of CD4+ PTCL-NOS; OR CD4+ AITL; OR CD4+ CTCL(either MF or SS).
4. Relapsed or refractory disease with at least two prior lines of systemic antineoplastic therapy.

   * Subjects with confirmed CD30+ PTCL or MF must have previously received brentuximab vedotin.
   * Subjects should have received at least two prior lines of standard of care therapies.
5. For Subjects with PTCL-NOS or AITL, at least one measurable lesion according to the International Working Group (IWG) Response Criteria.
6. For subjects with CTCL, disease stage IIB or higher based on TNMB system.
7. Subjects must have an identified hematopoietic stem cell transplant (HSCT) donor available prior to enrollment. HLA typing may be performed for source identification.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Adequate organ function.
10. Women of childbearing potential must have a negative pregnancy test at screening.
11. All Subject must agree to practice a highly effective method of contraception.
12. Women and men must agree not to donate eggs (ova, oocytes) or sperm, respectively, until at least 1 year after receiving a LB1901.

Exclusion Criteria:

1. Histologically confirmed CD8+ TCL - CD8 positivity in tumor must be confirmed within 3 months prior to apheresis by IHC or flow cytometry.
2. Prior treatment with cellular immunotherapy (e.g., CAR-T) or gene therapy product directed at any target.
3. Prior treatment with CD4-targeted therapy.
4. History of allogeneic haematopoietic stem cells transplant.
5. Antitumor therapy prior to apheresis as follows:

   * Any systemic anticancer therapy (chemotherapy, targeted therapy including ADC, epigenetic therapy including HDAC inhibitor, retinoids, pralatrexate, proteasome inhibitor therapy, investigational drug) within 21 days or at least 5 half-lives, whichever is shorter.
   * Anti-CCR4 monoclonal antibody or any other monoclonal antibody within 4 weeks or at least 5 half-lives, whichever is shorter.
   * Cytotoxic therapy within 14 days.
   * Immunomodulatory agent therapy within 7 days.
   * Radiotherapy within 14 days.
6. Immunosuppressant (e.g., cyclosporine or systemic steroids) above physiologic dosing within 7 days of apheresis.
7. Therapeutic anticoagulants (such as warfarin, heparin, low molecular weight heparin) (at least 3 half-lives must have elapsed after the last dose at the time of apheresis).
8. CNS disease prophylaxis (e.g., intrathecal methotrexate) at least 7 days before apheresis.
9. History or active Hepatitis B or C infection (except hepatitis C cured with pharmacotherapy); or history of or current HIV infection.
10. History of autoimmune disease requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.
11. Primary immunodeficiency.
12. Active CNS disease related to the underlying malignancy.
13. Stroke or seizure within 6 months of apheresis.
14. Impaired cardiac function or clinically significant cardiac disease.
15. Previous or concurrent malignancy with the following exceptions:

    * Adequately treated basal cell or squamous cell carcinoma.
    * In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to screening.
    * A primary malignancy which has been completely resected, or treated, and is in complete remission for at least 3 years prior to screening.
16. Serious and/or uncontrolled medical condition that, in the Investigator's judgment, would cause unacceptable safety risk.
17. Ongoing toxicity from previous anticancer therapy that has not resolved to baseline levels or to Grade 1 or less, except for alopecia, fatigue, nausea, and constipation.
18. Major surgery within 4 weeks prior to apheresis, or planned within 4 weeks after LB1901 administration.
19. Contraindications or life-threatening allergies, hypersensitivity, or intolerance to LB1901 or its excipients, including dimethyl sulfoxide; or to fludarabine, cyclophosphamide, or tocilizumab.
20. Contraindication or life-threatening allergy to valacyclovir, unless another suitable option of antiviral prophylaxis is identified after consultation with an Infectious Disease specialist.
21. Pregnant or breast-feeding.
22. Plans to become pregnant or breastfeed, or father a child within 1 year after receiving a LB1901 infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To characterize the safety and tolerability of LB1901 and determine the optimal dose or recommended dose for expansion (RDE). | Up to 2 years
  Multiple doses will be tested to establish a recommended dose.
To further characterize the safety and tolerability of LB1901 with the RDE identified in the dose escalation and determine the recommended Phase 2 dose (RP2D). | Up to 2 years
  Treatment of additional patients at the recommended dose as identified in the initial dose escalation part of the study.

SECONDARY OUTCOMES:
Over all Response | Up to 4 years
  Based on International Working Group Response Criteria for PTCL. Global Composite Response for CTCL
Time to response (TTR) | Up to 4 years
  Based on International Working Group Response Criteria for PTCL. Global Composite Response for CTCL
Duration of response (DOR) | Up to 4 years
  Based on International Working Group Response Criteria for PTCL. Global Composite Response for CTCL
Disease control rate (DCR) | Up to 4 years
  Based on International Working Group Response Criteria for PTCL. Global Composite Response for CTCL
Progression-free survival (PFS) | Up to 4 years
  Based on International Working Group Response Criteria for PTCL. Global Composite Response for CTCL
Overall survival (OS) | Up to 4 years
  Based on International Working Group Response Criteria for PTCL. Global Composite Response for CTCL

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Mayo Clinic, Rochester, Minnesota
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No